CLINICAL TRIAL: NCT06576414
Title: Feasibility, Effectiveness, and Patient Experience of Online Acceptance and Commitment Therapy Plus Exercises Versus Online Education Plus Exercises for Older People With Chronic Low Back Pain: A Pilot Randomized Controlled Trial
Brief Title: Feasibility, Effectiveness, and Patient Experience of Online Acceptance and Commitment Therapy Plus Exercises for Older People With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20240503001
Record Dates: First submitted 2024-05-13; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain (CLBP); Acceptance and commitment therapy (ACT); Psychological flexibility; Online intervention
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded (participants and statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older people with online ACT intervention (Experimental): 4 week ACT plus back exercise group
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: back exercise
- Older people without ACT intervention (Active Comparator): 4-week back exercise control group
  Interventions: Behavioral: back exercise; Behavioral: back care education

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — the first hour of ACT intervention followed by 1 hour of back exercise class, which led by a trained ACT counsellor and a trained exercise trainer
  Arms: Older people with online ACT intervention
Behavioral: back exercise — 1 hour of back exercise class led by a trained exercise trainer
Behavioral: back care education — 1 hour long interactive lesson to participants about LBP-related pathology, disability, psychology, and pain management skills.
  Arms: Older people without ACT intervention

SUMMARY:
No study has investigated the effects of online ACT on community-dwelling older adults. Given that clinical practice guidelines have recommended exercise therapy for treating people with CLBP, a combination of ACT and exercise therapy may yield better clinical outcomes than exercise alone among community-dwelling older adults with CLBP.

A double-blinded (participants and statistician) pilot randomized controlled trial (RCT) will be conducted to evaluate the feasibility and the relative effects of online ACT plus back exercise training as compared to exercise alone in improving psychological flexibility, physical well-being, and quality of life of community-dwelling older people with CLBP at different time points. The clinical outcomes will be measured at baseline, immediately after the 4-week treatment, and at the 3- and 6-month post-treatment follow-ups. Further, a qualitative research study will be conducted to understand the experiences of participating in online ACT and back exercise training in older people with CLBP (including identifying facilitators and barriers to participation).

DETAILED DESCRIPTION:
Recruitment posters will be displayed in five Hong Kong community centers. A total of 40 older people with LBP will be recruited and randomized to either a 4-week online ACT-plus-back-exercise group or a 4-week online spine care education-back-exercise control group. All participants will be screened for eligibility.

After providing the informed consent, participants will undergo baseline assessments. Then they will be randomized into either group. Immediately after the 4-week treatment and at 3- and 6-month post-treatment, participants will be invited to complete another set of questionnaires that are identical to their baseline questionnaires to evaluate the effects of interventions on their pain, physical function, psychological well-being, and quality of life.

Semi-structured interviews will be conducted to collect the user experience of participants in both groups by purposive sampling. The interviews will be conducted immediately post-treatment and at the 6-month post-treatment follow-up to evaluate the perspectives at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. have non-specific LBP in or near the lumbosacral spine with or without leg pain that lasts for at least 3-months in the last 12 months
2. have sought some medical or healthcare professional treatments for CLBP
3. able to read and write at an adequate level of proficiency in Chinese
4. Mini-Mental Status Examination (MMSE) scores 23 or above

Exclusion Criteria:

1. people with malignant pain or lumbar spinal stenosis
2. confirmed dementia
3. severe cognitive impairment
4. serious psychiatric or psychological disorders
5. Mini-Mental Status Examination (MMSE) scores below 23

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of psychological flexibility at immediately after the 4-week treatments | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment (All these time points are consistent with the description)
  The 7-item Chinese version of the Acceptance and Action Questionnaire II (AAQ-II) will be used to measure participants' psychological flexibility. It comprises 7 statements, which are rated on a 7-point scale, where 1 means "never true" and 7 means "always true." The maximum total score is 49. Higher total scores mean less flexibility. AAQII has been cross-culturally adapted and validated among local adolescents and has demonstrated satisfactory internal consistency and test-retest reliability.

SECONDARY OUTCOMES:
Change of LBP intensity | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment
  An 11-point numeric pain rating scale will be used to measure LBP intensity, where 0 means no pain and 10 means the worst imaginable pain. Participants need to report their back pain in the current moment, in the last 24 hours and the last 3 months.
Change of LBP-related disability | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment
  The Chinese version of 24-item Roland Morris Disability Index will be used to evaluate the LBP-related disability in older adults.30 It consists of 24 yes/no items related to LBP-related functional limitations. The summation of the scores of items with "yes" answer indicates the severity of LBP-related disability. The maximum score is 24.
Change of health-related quality of life | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment
  The Chinese version of EuroQol-5 Dimensions-levels (EQ-5D-5L) will be used to measure health-related quality of life (HRQOL) in our participants. It comprises 5 items related to mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each item has 5 options (no problem, slight problems, moderate problems, severe problems, extreme problems/unable to). It has been found to useful in monitoring HRQOL responses to treatment.
Change of depression, anxiety, and stress | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment
  The Chinese version of 21-item Depression, Anxiety Stress Scales (DASS) will be used to evaluate depression (7 items), anxiety (7 items), and stress (7 items) in older adults. Each item is rated on a 4-point scale ranging from 0 (not at all) to 3 (most of the time). Higher scores imply more mental health issues. It has been cross-culturally adapted to Hong Kong settings. DASS has demonstrated excellent internal consistency for depression, anxiety, and stress subscales.
Overall perceived changes in symptom severity, treatment response and the efficacy of treatment | Baseline, immediately after the 4-week treatment, and at 3- and 6-month post-treatment
  Global impression of change scale will be used to evaluate the overall perceived changes in symptom severity, treatment response and the efficacy of treatment immediately after the 4 week interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Arnold YL Wong, Hong Kong, None Selected, Hong Kong